CLINICAL TRIAL: NCT03160261
Title: Effect of Exenatide on Cortisol Secretion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Tartu (Other)
Responsible Party: Principal Investigator, Vallo Volke, Professor, University of Tartu
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Ex17
Record Dates: First submitted 2017-04-24; First posted 2017-05-19 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Healthy
MeSH Terms: interventions — Exenatide

STUDY DESIGN:
Intervention Model Description: Single-group, open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exenatide (Experimental): Single injection of 10 μg Exenatide subcutaneously.
  Interventions: Drug: Exenatide Injection

INTERVENTIONS:
Drug: Exenatide Injection — Single injection of Exenatide 10μg subcutaneously

SUMMARY:
The primary aim of the study is to describe the effect of single dose of 10 micrograms (μg) exenatide given subcutaneously (s/c) on cortisol secretion. Secondary outcomes involve ACTH and glucose levels.

DETAILED DESCRIPTION:
Exenatide is a short-acting Glucagon-Like Peptide receptor 1 (GLP-1 R) agonist.

The clinical trial is conducted in10 healthy volunteers. Each subject receives one dose of subcutaneous exenatide (10 μg). After that, hormonal and physiological changes are measured during two hours. The blood samples are taken in 30-minute intervals.

The primary endpoint is peak value of cortisol achieved during the 2 hours after drug administration.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years
* Body weight >65 kg

Exclusion Criteria:

* Presence of chronic illness
* daily use of any medicines
* pregnancy, lactation
* use of oral contraceptives during previous 2 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2017-12-28 (Actual); Study Completion 2017-12-28 (Actual)

PRIMARY OUTCOMES:
Cortisol peak | every 30 minutes during 2 hours after injection
  Maximum concentration achieved after exenatide dose (any timepoint after injection)

SECONDARY OUTCOMES:
Adrenocorticotropin (ACTH) peak | every 30 minutes during 2 hours after injection
  Maximum concentration achieved after exenatide dose (any timepoint after injection)
Glucose | Glucose measured every 30 minutes during 2 hours after injection
  Glucose values' area under the curve
Growth hormone | every 30 minutes during 2 hours after injection
  Maximum concentration achieved after exenatide dose (any timepoint after injection)

OTHER OUTCOMES:
heart rate | every 30 minutes during 2 hours after injection
  Change in heart rate
Blood pressure | every 30 minutes during 2 hours after injection
  Change in blood pressure
nausea | every 30 minutes during 2 hours after injection
  intensity of nausea in visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Vallo Volke, MD,PhD, Principal Investigator — University of Tartu
Locations (1):
- Tartu University Hospital, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heinla K, Vasar E, Reppo I, Sedman T, Volke V. GLP-1 Receptor Agonists Induce Growth Hormone Secretion in Healthy Volunteers. Diabetes Ther. 2023 Apr;14(4):777-786. doi: 10.1007/s13300-023-01381-w. Epub 2023 Feb 17. PMID 36800161